CLINICAL TRIAL: NCT04165642
Title: Single-Laser PVI: Single-encirclement Laserballoon Ablation for Pulmonary Veins Isolation
Acronym: SingleLaser
Status: Terminated | Type: Observational
Why Stopped: due to unattainability of the expected sampling unit.
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Chief of the Department of Arrhythmology and Electrophysiology, IRCCS Policlinico S. Donato
Other Study IDs: Paroxysmal or persistent AF
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Assessment of Safety of Laser Balloon Ablation; Assessment of Procedural Times of Laser Ballon Ablation
Keywords: laser ballon ablation; laser ballon; pulmonary vein isolation; atrial fibrillation; AF ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Laser ballon ablation for Pulmonary vein isolation — The patients indicated to AF ablation procedure will be treated with laser balloon ablation without verification of electrical isolation of pulmonary veins using implantable loop recorder and/or Holter monitoring

SUMMARY:
To assess the efficacy of laser balloon ablation of atrial fibrillation (AF) without verification of electrical isolation of pulmonary veins using implantable loop recorder.

This is a prospective and single-center study. A targeted number of 82 patients suffering from paroxysmal or persistent AF, indicated to undergo catheter ablation will be included. The study will consist of: i) patient enrolment, ii) treatment phase, and iii) 1-year follow-up phase. The duration of the study is expected to be 24 months, from first patient enrolment to last patient follow up.

DETAILED DESCRIPTION:
This is a prospective and single-center study. A targeted number of 82 patients suffering from paroxysmal or persistent AF, indicated to undergo catheter ablation will be included. The study will consist of: i) patient enrolment, ii) treatment phase, and iii) 1-year follow-up phase. The duration of the study is expected to be 24 months, from first patient enrolment to last patient follow up.

In a recent meta-analysis including 1188 patients, free from arrhythmic recurrences at 12 months after a single ablative procedure with a laser balloon and without continuous monitoring with ILR was 74%1.

Assuming that the approach without post-ablative verification of pulmonary vein isolation and continuous monitoring with ILR can lead to a 60% success rate at 12 months, 80 patients are required to have an 80% probability to observe a level of 2-code significance of 0.05 in an exponential model with the log rank test. With an estimated loss of data (patients lost to follow-up, protocol deviations and incomplete data) of 5%, the total number of patients to be enrolled is 82.

Subject screening and enrolment will be carried out for approximately 12 months. The study will continue up to 12 months after last patient enrolment, dependent on the rate of enrolment and the regulatory timeline (as applicable).

ELIGIBILITY:
Inclusion Criteria:

To participate in this clinical subject, the subject must meet all of the following inclusion criteria:

* Age between 18 and 85 years
* Paroxysmal or persistent AF
* Patients AF who have indications for the first time ablation procedure according to the ESC / EHRA recommendations (European Society of Cardiology / European Heart Rhythm Association).
* Ability to provide written informed consent for study participation and be willing and able to comply with the study evaluations and follow up schedule

Exclusion Criteria:

Subjects are not eligible for clinical study participation if they meet any of the following exclusion criteria:

* Previous AF ablation procedures
* Secondary AF due to other causes
* Hyperthyroidism
* Left ventricular ejection fraction <30%
* NYHA class IV
* Left atrium area > 35 cm2
* Severe disease of cardiac valves
* Contraindication to anticoagulant therapy
* Presence of thrombus in the left atrium
* Myocardial infarction or unstable angina or recent coronary artery bypass (<6 months)
* Thoracic surgery for congenital, valvular or aortic disease
* History of cerebrovascular events
* Pregnancy
* Significant comorbidity, such as cancer, severe kidney failure requiring dialysis, severe obstructive pulmonary disease, cirrhosis, with a life expectancy of less than 2 years
* Contraindications are present as indicated in the "instructions for use" of the devices used

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients referred to the Department of Arrhythmology for the management of parosysmal or persistent AF will be considered for eligibility. A subject, who meets all of the inclusion criteria, and none of the exclusion criteria, is eligible to participate in this study. All subjects enrolled in the clinical study (including those withdrawn from the clinical study or lost to follow-up) will be accounted for and documented, assigning an identification code linked to their names, alternative identification or contact information.
  This log will be kept up to date throughout the clinical study by the principal investigator (PI) or his/her authorized designee. To ensure subject privacy and confidentiality of data this log must be maintained throughout the clinical study at the clinical site.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Success rate at 1 year | 12 months after ablation
  Free from AF, atrial tachycardia and flutter documented with ILR or Holter ECG monitorwithout antiarrhythmic drugs.

SECONDARY OUTCOMES:
Procedural and 1-year complications related to the ablation procedure. | during the procedure and 12 months after ablation
  Procedural and 1-year complications related to the ablation procedure.
inducibility of AF after the procedures | During the procedure
  programmed atrial stimulation before and after isoproterenol
AF Burden | 12 months after ablation
  Assessment of AF burden by holter monitoring or implantable loop recorder

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, PhD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT04165642/Prot_000.pdf